CLINICAL TRIAL: NCT04021784
Title: Limited-efficacy Testing of Spring Distraction System (SDS) and a Bilateral One Way Rod (NEMOST) for Early Onset Neuromuscular Scoliosis (BiPOWR)
Brief Title: Limited-efficacy Testing of SDS and NEMOST for Early Onset Neuromuscular Scoliosis
Acronym: BiPOWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: EUROS (Industry)
Responsible Party: Principal Investigator, M.C. Kruyt, MD, PhD, Orthopaedic surgeon, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL 64018.041.17
Record Dates: First submitted 2019-06-13; First posted 2019-07-16 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Neuromuscular Scoliosis; Distraction System; Growth Friendly System

STUDY DESIGN:
Intervention Model Description: Half of the patients will be implanted with SDS system, the other half will be implanted with NEMOST.
Who Masked: Participant
Masking Description: The patient is blinded to the medical device until after surgery. This is done to prevent selection bias through withdrawal. Patients are unblinded post-operatively, to enable accurate patient counseling with radiographs, on which the implant can be clearly seen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spring Distraction System (SDS) (Experimental): The SDS will be placed and fits around a standard rod of 5.5mm.
  Interventions: Device: SDS
- Necker Enfants Malade OSTeosynthesis (NEMOST) (Experimental): The NEMOST is a one-way-rod that uses a ratchet type of locking mechanism. Both NEMOST devices should be placed in parallel, on the two fixator rods that are connected with a cross connector
  Interventions: Device: NEMOST

INTERVENTIONS:
Device: SDS — The patient is implanted with SDS.
  Arms: Spring Distraction System (SDS)
Device: NEMOST — The patient is implanted with NEMOST.
  Arms: Necker Enfants Malade OSTeosynthesis (NEMOST)

SUMMARY:
The primary aim of this study is to investigate and describe the limited efficacy of the Spring Distraction System (SDS) and Bilateral One Way Rod (NEMOST) in maintaining curve reduction without repeat lengthening procedures and complications.

Secondary aims are to describe growth of the instrumented spine, health-related quality of life, and to compare both devices.

DETAILED DESCRIPTION:
Several innovative solutions have been developed to treat growing children with a severe scoliosis. One device (SDS) was developed internally at the department of orthopaedics UMC Utrecht in the Netherlands. The other device (NEMOST) was developed at the Necker Hospital in France.

This study is designed as a multicenter, limited-efficacy study using two prospective cohorts according a randomised clinical trial. The study will be performed in two centers (UMC Utrecht, Amsterdam UMC and Erasmus MC).

Primary endpoints are the limited-efficacy in terms of maintenance of curve correction and occurrence of SAEs related to the procedure. These data will be compared to a recently described cohort of patients that received a "standard treatment", the MGCR (Skov et al., 2017). Secondary endpoints include spinal- and implant growth, patient performance based on the EOSQ 24 questionnaire and surgical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Non ambulant
* Neuromuscular or syndromal scoliosis
* Progressive scoliosis indicated for bipolar fixation extending to the pelvis
* Diagnosis of scoliosis before age 10
* Patient under 12 and open triradiate cartilage (usually closes around 12 years for girls and 14 years for boys)
* Main curve proximal end vertebra below Th 3
* Non rigid curve
* Patients who have an indication for a primary surgery

Exclusion Criteria:

* Ambulant
* Patients with closed triradiate cartilage
* Patients with a skeletal dysplasia that effects growth (Achondroplasia, SED)
* Patients with a systemic disease which severely influences bone quality e.g. osteogenesis imperfecta, metabolic diseases
* Patients with soft tissue weakness (Ehler Danlos, Marfan, Neurofibromatosis, Prader Willi)
* Patients that have a congenital anomaly of the spine of more than 5 vertebrae
* Patients with an active systemic disease such as JIA, HIV, oncologic treatment
* Patients with a previous surgical fusion of the spine
* Patients that are expected to be lost to FU due to e.g. likely to immigrate within 1 year.
* Patients that have had a previous spine surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Limited-efficacy of SDS and NEMOST in terms of curve correction maintenance | Until 1 year post-operatively
  Changes in cobb angle on radiographs post-op and at 4 weeks, 3 months, 6 months and 12 months follow-up (FU). A maximum of 5 degrees increase will be the threshold to define maintenance.
Incidence of possible Treatment-Emergent Serious Adverse Events of SDS and NEMOST | Until 1 year post-operatively
  Reported treatment related Serious Adverse Events (SAEs) per-operatively and at 4 weeks, 3 months, 6 months and 12 months FU.

SECONDARY OUTCOMES:
Limited-efficacy of SDS and NEMOST in terms of spinal length | Until 1 year post-operatively
  Changes in length of T1-T12, T1-S1 and the instrumented segment in mm on calibrated Anterior Posterior (AP) X-rays post-op and at 4 weeks, 3 months, 6 months and 12 months FU.
SDS vs. NEMOST with respect to limited-efficacy in terms of curve correction maintenance | Until 1 year post-operatively
  Changes in cobb angle on radiographs post-op and at 4 weeks, 3 months, 6 months and 12 months follow-up (FU). A maximum of 5 degrees increase will be the threshold to define maintenance.
SDS vs. NEMOST with respect to limited-efficacy in terms of spinal length | Until 1 year post-operatively
  Changes in length of T1-T12, T1-S1 and the instrumented segment in mm on calibrated AP X-rays post-op and at 4 weeks, 3 months, 6 months and 12 months FU.
SDS vs. NEMOST with respect to the development of the sagittale profile and instrumented thoracic kyphosis | Until 1 year post-operatively
  Changes in sagittal profile and thoracic kyphosis and the instrumented (T1 pelvic angle, TPA) segment in mm on calibrated Anterior Posterior (AP) X-rays post-op and at 4 weeks, 3 months, 6 months and 12 months FU.
SDS vs. NEMOST with respect to surgery time | Until 1 year post-operatively
  Surgery time in minutes
SDS vs. NEMOST with respect to blood loss during surgery | Until 1 year post-operatively
  Blood loss in cc
SDS vs. NEMOST with respect to length of hospital stay | Until 1 year post-operatively
  Length of hospital stay in days
SDS vs. NEMOST with respect to recovery time | Until 1 year post-operatively
  Recovery time in minutes
SDS vs. NEMOST with respect to the incidence of disease- or treatment-related Serious Adverse Events | Until 1 year post-operatively
  Reported treatment related SAEs per-operatively and at 4 weeks, 3 months, 6 months and 12 months FU.
SDS vs. NEMOST with respect to 3D development of the spine | Pre-operatively
  Apical Vertebral Rotation based on bone MRI
SDS vs. NEMOST with respect to Quality Of Life (QOL) on the Early Onset Scoliosis Questionnaires (EOSQ-24) | Until 1 year post-operatively
  Parent reported QOL and performance is assessed with the 24-item Early Onset Scoliosis Questionnaires (EOSQ-24) pre-op and at 4 weeks, 3 months, 6 months and 12 months FU. EOSQ-24 covers the following domains: Child's Health Related Quality of Life (16 items), Family Impact (2 items) and Satisfaction (2 items).
SDS vs. NEMOST with respect to the effect on the development of the pelvic obliquity | Until 1 year post-operatively
  Changes in pelvic obliquity on X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Moyo C Kruyt, MD, PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemans JVC, Tabeling CS, Scholten EP, Stempels HW, Miladi L, Castelein RM, Kruyt MC. Surgical treatment of neuromuscular Early Onset Scoliosis with a bilateral posterior one-way rod compared to the Spring Distraction System: study protocol for a limited-efficacy Randomized Controlled Trial (BiPOWR). BMC Musculoskelet Disord. 2023 Jan 10;24(1):20. doi: 10.1186/s12891-022-06048-4. PMID 36627616
- See also: Surgical treatment of neuromuscular Early Onset Scoliosis with a bilateral posterior one-way rod compared to the Spring Distraction System: study protocol for a limited-efficacy Randomized Controlled Trial (BiPOWR) — https://link.springer.com/article/10.1186/s12891-022-06048-4